CLINICAL TRIAL: NCT00010244
Title: Conformational, Curative Ratiotherapy For Prostate Cancer (NO, N-): Phase III Multicenter Study Of The Contribution To Survival Without Clinical Or Biological Change With A Dose Variation Of 15% (80 Gy VS 70 Gy)
Brief Title: Comparison of Radiation Therapy Regimens in Treating Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0160/9901; FRE-FNCLCC-PAC-GETUG-06-99001 (Other: UNICANCER); EU-20037 (Registry Identifier: European Union)
Record Dates: First submitted 2001-02-02; First posted 2004-02-04 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known which regimen of radiation therapy is more effective for prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of different regimens of radiation therapy in treating patients who have localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the 5-year survival rate, in terms of clinical and biological remission, in patients with localized prostate cancer treated with two different radiotherapy regimens using different doses and number of fractions. II. Compare the nadir of PSA and the delay in obtaining the nadir in patients treated with these two regimens. III. Compare acute and long-term toxicity of these two regimens in these patients. IV. Compare overall survival and quality of life in patients treated with these two regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms. Arm I: Patients receive radiotherapy to the seminal vesicles at 46 Gy in 23 fractions and to the prostate at 70 Gy in 35 fractions, with 5 fractions per week. Arm II: Patients receive radiotherapy to the seminal vesicles as in arm I and to the prostate at 80 Gy in 40 fractions, with 5 fractions per week. Treatment continues in both arms in the absence of disease progression or unacceptable toxicity. Quality of life is assessed annually. Patients are followed every 4 months for a minimum of 5 years.

PROJECTED ACCRUAL: A total of 306 patients (153 per arm) will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Localized prostate cancer: T2a-T3a OR T1b or T1c with PSA at least 10 ng/mL OR T1b or T1c with Gleason score 7-10 No T3b or T4; positive biopsy of nodal excision N0, or any N with bilateral removal and the estimated risk of nodal invasion is at least 10% M0 (by bone scintograph and chest x-ray) PSA less than 50 ng/mL

PATIENT CHARACTERISTICS: Age: Under 75 Performance status: WHO 0-1 Life expectancy: At least 10 years Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No other prior invasive malignancy within the past 5 years except basal cell carcinoma No social, familial, or geographic obstacles that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy No concurrent biologic therapy Chemotherapy: No prior chemotherapy No concurrent chemotherapy Endocrine therapy: No prior hormonal therapy including adjuvant therapy No concurrent hormonal therapy Radiotherapy: No prior pelvic radiotherapy Surgery: No prior radical anterior prostatectomy for cancer No prior castration

Ages: 0 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 1999-09 (Actual); Primary Completion 2007-02-20 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: V. Beckendorf, MD, Study Chair — Centre Alexis Vautrin
Locations (19):
- France (19):
  - Hopital Saint Andre, Bordeaux
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - Institut Curie - Section Medicale, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Jules Courmont - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Jean Bernard, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Beckendorf V, Guerif S, Le Prise E, Cosset JM, Bougnoux A, Chauvet B, Salem N, Chapet O, Bourdain S, Bachaud JM, Maingon P, Hannoun-Levi JM, Malissard L, Simon JM, Pommier P, Hay M, Dubray B, Lagrange JL, Luporsi E, Bey P. 70 Gy versus 80 Gy in localized prostate cancer: 5-year results of GETUG 06 randomized trial. Int J Radiat Oncol Biol Phys. 2011 Jul 15;80(4):1056-63. doi: 10.1016/j.ijrobp.2010.03.049. Epub 2010 Dec 14. PMID 21147514
- [Derived] Kim S, Kong JH, Lee Y, Lee JY, Kang TW, Kong TH, Kim MH, You SH. Dose-escalated radiotherapy for clinically localized and locally advanced prostate cancer. Cochrane Database Syst Rev. 2023 Mar 8;3(3):CD012817. doi: 10.1002/14651858.CD012817.pub2. PMID 36884035